CLINICAL TRIAL: NCT07219485
Title: An Open-Label Study to Evaluate Safety of Pitolisant in Participants With Prader-Willi Syndrome
Brief Title: A Study of Pitolisant in Participants With Prader-Willi Syndrome
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Harmony Biosciences Management, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBS-101-CL-314
Record Dates: First submitted 2025-10-20; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Prader-Willi Syndrome
Keywords: Pitolisant; HBS-101; Prader-Willi syndrome; PWS
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — pitolisant

STUDY DESIGN:
Intervention Model Description: All participants receive pitolisant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pitolisant (Experimental): All participants receive pitolisant administered orally once daily in the morning upon awakening.
  Interventions: Drug: Pitolisant

INTERVENTIONS:
Drug: Pitolisant — * Pitolisant 4.45 mg tablets
  * Pitolisant 17.8 mg tablets
  Other Names: HBS-101

SUMMARY:
The purpose of this study is to assess safety of pitolisant in eligible participants with Prader-Willi syndrome (PWS) who completed the End of Treatment (EOT) visit in a parent study (HBS-101-CL-002 [Open Label Extension (OLE)], HBS- 101-CL-004, or HBS-101-CL-312 OLE).

DETAILED DESCRIPTION:
This is a Phase 3, open-label study evaluating the long-term safety of pitolisant in approximately 150 participants with Prader-Willi syndrome who have completed participation in qualifying parent studies (HBS-101-CL-002 [OLE], HBS-101-CL-004, or HBS-101-CL-312 [OLE]).

Safety assessments will be conducted every 6 months. This study is open to participants from the qualified parent studies who were enrolled at US sites only.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet the following criteria to be enrolled in this study:

1. Ability to provide voluntary, written informed consent (participant, if applicable, or parent[s]/legal guardian[s]) and, where applicable, voluntary, written assent (participant, as appropriate).
2. Completion of an EOT visit in one of the following parent studies with pitolisant: HBS-101-CL-002 (OLE), HBS-101-CL-004, or HBS-101-CL-312 (OLE).

   Note: The parent study EOT visit may be completed after the participant completes screening for study HBS-101-CL-314 to allow for continuation of study drug between the 2 studies.
3. A participant who is a female of childbearing potential (FCBP) must have a negative urine pregnancy test at the last in-person visit of the parent study prior to screening and must agree to remain abstinent or use an effective method of nonhormonal contraception to prevent pregnancy for the duration of the study and for 21 days after final dose of study drug. Participants using hormonal contraception must also use an alternative nonhormonal contraceptive method during treatment with pitolisant and for at least 21 days after discontinuing treatment. An FCBP is defined as a female who is post menarche, has an intact uterus and at least 1 ovary, and is <1 year postmenopausal.
4. Male participants who are not azoospermic (vasectomized or due to a medical cause) must agree to use a barrier method of contraception for the duration of the study and for 21 days after the final dose of study drug.
5. In the opinion of the Investigator, the participant/parent(s)/legal guardian(s) are capable of understanding and willing to comply with the requirements of the protocol and administration of oral study drug.

Exclusion Criteria:

A participant who meets any of the following criteria will be excluded from enrollment in the study:

1. Does not agree to discontinue any prohibited medication or substances listed in this protocol.
2. Is planning to breastfeed over the course of the study. Lactating women must agree not to breastfeed for the duration of the study and for 7 days after final dose of study drug.
3. Participation in an interventional research study with an investigational medication or device, other than pitolisant, for the duration of the study.
4. Has a body surface area (BSA) corrected estimated glomerular filtration rate (eGFR) of <15 mL/minute.
5. Has a history of severe hepatic impairment (Child-Pugh Class C).
6. Is receiving or is unable to discontinue a medication known to prolong the QT interval.
7. Has a significant risk of committing suicide or suicidality based on history, routine psychiatric examination, Investigator's judgment, or an answer of "yes" to question 4 or 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS), that was completed at the last visit in the parent study.
8. Based on the judgment of the Investigator, is unsuitable for the study for any reason, including but not limited to unstable or uncontrolled medical conditions (including psychiatric and neurological conditions) or a medical condition that might interfere with the conduct of the study, confound interpretation of study results, pose a health risk to the participant, or compromise the integrity of the study.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants reporting Treatment-Emergent Adverse Events (TEAEs) | From the end of the EOT visit of the parent study through 30 days after the final dose of study drug.
  A treatment-emergent adverse event (TEAE) is any adverse event reported during treatment with study drug in this study and up to 30 days after final dose of study drug, or any worsening of a pre-existing condition reported during treatment with study drug and up to 30 days after final dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: David Seiden, MD, Study Director — Harmony Biosciences Management, Inc.
Locations (1):
- Science 37, Morrisville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No